CLINICAL TRIAL: NCT02173314
Title: Permanency Innovations Initiative- Nevada Initiative to Reduce Long-Term Foster Care
Brief Title: Nevada Initiative to Reduce Long-Term Foster Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 8977-2
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: At Risk for Foster; In Foster Care
Keywords: Long term foster care; child abuse and neglect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: SAFE FC
- Comparison (No Intervention)

INTERVENTIONS:
Other: SAFE FC — SAFE - FC, a combination of SAFE (developed by ACTION for Child Protection) and Family Connections (developed by Ruth H. Young Center for Families and Children, University of Maryland School of Social Work) for Populations 1 and 2.
  Other Names: SAFE - FC, a combination of SAFE and Family Connections
  Arms: Treatment

SUMMARY:
The evaluation of the Nevada Initiative to Reduce Long-Term Foster Care (LTFC) includes three populations. It will examine how the interventions SAFE- FC and FSE impact or relate to permanency outcomes for children most at risk for long term foster care and currently in care.

DETAILED DESCRIPTION:
The project targets three populations of children. For populations 1 and 2, the study will evaluate an intervention known as SAFE-FC. The intervention aims to prevent long term foster care by providing tailored services and intensive engagement with all new families with children identified as unsafe (Population 1) and for cases that are currently in care and at risk of LTFC where reunification is the case goal (Population 2). Family Search and Engagement (FSE) is the intervention for Population 3; it involves intense search practices to identify possible permanency resources. For Populations 1 and 2 the study is a randomized, intent-to-treat design to measure safety and permanency outcomes. For Population 3 the evaluation will be a descriptive study to analyze relationships between the intervention approach and outcomes. Both studies aim to examine how the interventions (SAFE- FC and FSE) impact or relate to permanency outcomes for children most at risk for long term foster care.

ELIGIBILITY:
Inclusion Criteria:

* Children assessed to be unsafe via the Nevada Initial Assessment
* children in foster care with specific risk characteristics.

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 507 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to stable permanence | Measured from the date of random assignment to the discharge date or to the end of the study period for cases that did not discharge
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS)
Caregiver readiness for change | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Measured with Readiness for Parenting Change Scale (REDI) Abbreviated (Chaffin et al, 2011)

SECONDARY OUTCOMES:
Caregiver stress | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Parenting Stress Index - Short Form (PSI-SF) (Abidin, 1983)

OTHER OUTCOMES:
Caregiver mental health | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Brief Symptoms Inventory (BSI) (Derogatis, 1993)
Child behavior/mental health problems | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Child Behavior Checklist (CBCL) (Achenbach, 1991)
Positive parenting attitudes | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Adult-Adolescent Parenting Inventory (AAPI-2) (Bavolek & Keene, 1999)
Social support | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Social Provisions Scale (SPS) (Russell & Cutrona, 1984)
Helping alliance for both caregiver and worker | Measured at 6 months and again at case closure (duration of their involvement with Washoe County DSS is on average 24 months)
  Helping Relationship Inventory (Poulin & Young, 1997)
Resiliency | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Resiliency Attitudes Scale (RAS) (Briscoe, B. & Harris, B., 1994)
Home stability | Measured at intake, at 6 months, 12 months, 18 months, and again at case closure (participants will be followed throughout the duration of their involvement with Washoe County DSS which is on average 24 months)
  Based on subscales of the CWBS (questions from Zuravin & DePanfilis, 1996)
Time to permanency | Measured every six months in calendar year
  State administrative data system
Recurrence of child abuse and neglect | Measured every six months in calendar year
  State administrative data system
Placement rate (population 1 only) | Measured every six months in calendar year
  State administrative data system
Time for case closure | Measured every six months in calendar year
  State administrative data system
Time to reunification | Measured every six months in calendar year
  State administrative data system
Foster care re entry rate | Measured every six months in calendar year
  State administrative data system

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sedlak, PhD., Study Director — Westat; Mark Testa, PhD., Principal Investigator — University of North Carolina